CLINICAL TRIAL: NCT02216968
Title: Increasing Vegetable Intake in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Theresa A Nicklas, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: H-30554; 1R21HD073608-01A1 (NIH)
Record Dates: First submitted 2014-08-06; First posted 2014-08-15 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Obesity; Behavior; Food Habits
Keywords: vegetables; Head Start; preschool; children; theater; puppet
MeSH Terms: conditions — Obesity; Behavior; Feeding Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AA - Increase vegetable intake (Experimental): 60 African-American (AA) preschool children will participate in the Intervention Group. 60 AA children will belong to the Control Group.
  6-week Intervention: 120 AA and HA children will be shown the Puppet Shows and will be given a bag of ingredients to prepare the vegetable highlighted that week in the Puppet Show. The 6 week intervention includes a baseline assessment (1 week), followed by the intervention (4 weeks), and post assessment (1 week). The primary hypothesis to be tested is children who receive the PUPPET intervention with a parent/teacher component will demonstrate "increase vegetable intake in pre-school children".
  Interventions: Behavioral: Increase vegetable intake in pre-school children
- HA - Increase vegetable intake (Experimental): 60 Hispanic-American (HA) preschool children will participate in the Intervention Group. 60 HA children will belong to the Control Group.
  6-week Intervention: 120 AA and HA children will be shown the Puppet Shows and will be given a bag of ingredients to prepare the vegetable highlighted that week in the Puppet Show. The 6 week intervention includes a baseline assessment (1 week), followed by the intervention (4 weeks), and post assessment (1 week). The primary hypothesis to be tested is children who receive the PUPPET intervention with a parent/teacher component will demonstrate "increase vegetable intake in pre-school children".
  Interventions: Behavioral: Increase vegetable intake in pre-school children

INTERVENTIONS:
Behavioral: Increase vegetable intake in pre-school children — 6-week Intervention: 120 AA and HA children will be shown the Puppet Shows and will be given a bag of ingredients to prepare the vegetable highlighted that week in the Puppet Show. The 6 week intervention includes a baseline assessment (1 week), followed by the intervention (4 weeks), and post assessment (1 week). The primary hypothesis to be tested is children who receive the PUPPET intervention with a parent/teacher component will demonstrate "increase vegetable intake in pre-school children".

SUMMARY:
The purpose of this study is to test the feasibility of an innovative approach to increase the amount of vegetable's (V) intake consumed by preschool children who are predominately African-American (AA) and Hispanic-American (HA).

DETAILED DESCRIPTION:
The purpose of this study is to test the feasibility of an innovative approach to increase the amount of vegetable's (V) intake consumed by preschool children who are predominately African-American (AA) and Hispanic-American (HA).The primary endpoint will be changes in V consumption in high school children with the hypothesis that a puppet intervention will increase their V consumption by preschool children. To achieve the project goal, our specific aims (SA) are to: SA1: Successfully recruit 6 preschool (PS) centers and 168 AA and 168 HA children 3 to 5 y enrolled there. SA2: Conduct individual interviews for formative assessment of the PUPPET shows. SA3: Develop the manual of operation and intervention protocols SA4: Develop 4 videotaped theatre-based PUPPET shows that are developmentally and cognitively appropriate for use with 3- to 5-year-old AA and HA children SA5: Pilot-test the feasibility of the PUPPET intervention with 3 intervention and 3 control HS centers. SA6: Use the data collected in Aim 5 to estimate parameters required to conduct a group randomized trial for an evaluation of the efficacy of the intervention. The primary hypothesis (H1) to be tested is that children who receive the PUPPET intervention will demonstrate increased V consumption in HS compared to children in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* non-patient
* normals
* African-american
* Hispanic-american
* 3 to 5 y olds

Exclusion Criteria:

* pregnant woman
* neonates
* dietary restrictions
* chronic disease
* developmental disabilities
* special education
* does not read or write in spanish or english

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2012-07 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Vegetable Intake in Preschool Children | 1 year 11 months
  There will be 2 phases to program development: diagnostic and formative. The diagnostic phase will consist of 20 individual interviews with child-care providers and parents (½ AA, ½ HA) and 20 interviews with preschool children (½ AA, ½ HA).In addition the parents will be asked to complete the Cooking Confidence Questionnaire, the Barriers and Facilitators Questionnaire on Vegetables and a list of their child's favorite vegetables before coming to the interview. Implementation will include the showing of the 4 video-taped puppet shows to 10-12 children immediately prior to the lunch meal on 4 consecutive days. These children will be assessed at lunch using the digital diet estimation method.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa A Nicklas, DrPH, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Derived] Nicklas T, Lopez S, Liu Y, Saab R, Reiher R. Motivational theater to increase consumption of vegetable dishes by preschool children. Int J Behav Nutr Phys Act. 2017 Feb 7;14(1):16. doi: 10.1186/s12966-017-0468-0. PMID 28166788